CLINICAL TRIAL: NCT00802035
Title: A Phase 1, Single-Center, Open-Label Study of the Pharmacokinetics of Baclofen Formulations Administered to Healthy Adults
Brief Title: ALK29-002: A Study of Baclofen Formulations in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALK29-002
Record Dates: First submitted 2008-11-26; First posted 2008-12-04 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Alcohol Dependence
Keywords: ALK29; Alcohol Dependence; Pharmacokinetics
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IR am (Active Comparator): 30 mg, single dose, morning administration (immediate release [IR])
  Interventions: Drug: Baclofen IR
- ER am (Experimental): 30 mg; single dose; morning administration (extended release [ER])
  Interventions: Drug: Baclofen ER
- ER pm (Experimental): 30 mg; single dose; evening administration
  Interventions: Drug: Baclofen ER
- IR pm (Active Comparator): 30 mg; single dose; evening administration
  Interventions: Drug: Baclofen IR

INTERVENTIONS:
Drug: Baclofen IR — 30 mg; single dose
  Arms: IR am; IR pm
Drug: Baclofen ER — 30 mg; single dose
  Arms: ER am; ER pm

SUMMARY:
The purpose of this study is to determine the pharmacokinetics, safety, and tolerability of different baclofen formulations.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years
* Body mass index of 19 to 30 kg/m2 at screening
* If subject is female and of childbearing potential, she must agree to use an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* Pregnancy and/or currently breastfeeding
* Clinical significant medical condition or observed abnormalities
* Acute gastrointestinal disorder or history of chronic gastrointestinal disease or surgery
* Participation in a clinical trial within 30 days before screening
* Known intolerance and/or hypersensitivity to baclofen or its excipients
* Use of alcohol-, caffeine-, or xanthine-containing products
* Clinically significant illness within 30 days of first study drug administration
* Dietary restrictions that conflict with required study meals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 5 weeks

SECONDARY OUTCOMES:
Time to Cmax | 5 weeks
Significant abnormal laboratory findings | 5 weeks
Area under the plasma concentration curve (AUC) | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A. Bieberdorf, MD, CPI, Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States